CLINICAL TRIAL: NCT03247400
Title: The Evaluation of Vitiligous Lesions Repigmentation After the Administration of Atorvastatin Calcium Salt and Simvastatin-acid Sodium Salt in Patients With Active Vitiligo (EVRAAS)
Brief Title: The Evaluation of Vitiligous Lesions Repigmentation After the Administration of Atorvastatin Calcium Salt and Simvastatin-acid Sodium Salt in Patients With Active Vitiligo
Acronym: EVRAAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Rafal Czajkowski, Clinical Professor, Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCU 631
Record Dates: First submitted 2017-08-05; First posted 2017-08-11 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Non-segmental Vitiligo
MeSH Terms: interventions — Simvastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1% simvastatin-acid sodium salt ointment (Active Comparator): 1% simvastatin-acid sodium salt ointment applied onto a predefined limb compared with placebo ointment applied onto an opposite limb
  Interventions: Drug: 1% simvastatin-acid sodium salt ointment
- 1% atorvastatin calcium salt ointment (Active Comparator): 1% atorvastatin calcium salt ointment applied onto a predefined limb compared with placebo ointment applied onto an opposite limb
  Interventions: Drug: 1% atorvastatin calcium salt ointment
- Vehicle ointment (Placebo Comparator): Placebo ointment applied onto limbs opposite to treated with active substances
  Interventions: Drug: 1% simvastatin-acid sodium salt ointment; Drug: 1% atorvastatin calcium salt ointment

INTERVENTIONS:
Drug: 1% simvastatin-acid sodium salt ointment — 1% simvastatin-acid sodium salt ointment applied onto a predefined limb
  Other Names: simvastatin
  Arms: 1% simvastatin-acid sodium salt ointment; Vehicle ointment
Drug: 1% atorvastatin calcium salt ointment — 1% atorvastatin calcium salt ointment applied onto a predefined limb
  Other Names: atorvastatin
  Arms: 1% atorvastatin calcium salt ointment; Vehicle ointment

SUMMARY:
The aim of this study is to evaluate the influence of simvastatin and atorvastatin on vitiligous lesions in patients with non-segmental vitiligo.

DETAILED DESCRIPTION:
According to available data, statins act through several immunological pathways, potentially reversing undesirable phenomena underlying autoimmune vitiligo pathogenesis. A study has been designed as a single-center, randomized, double-blind, placebo-controlled pilot study with the enrollment of at least 20 active non-segmental vitiligo patients presenting with vitiligous lesions on both upper and lower limbs. Clinical effects of ointments containing 1% simvastatin-acid sodium salt or 1% atorvastatin calcium salt applied on a preselected limb will be assessed in comparison with vehicle ointment applied on the opposite limb. All study participants will undergo clinical evaluation using Body Surface Area (BSA) and Vitiligo Area Scoring Index (VASI) scales at baseline, week 4, week 8 and week 12 time points. Precise assessment of skin lesions will be performed using photographic documentation obtained during each study visit and processed with NIS-Elements software.

ELIGIBILITY:
Inclusion Criteria:

1. patients of Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University, Collegium Medicum in Bydgoszcz
2. provision of an informed consent form prior to any study procedures
3. diagnosis of non-segmental acrofacial vitiligo with upper and lower limbs involvement
4. active vitiligo, defined as appearance of new areas of depigmentation or progression of existing areas of depigmentation within 3 months preceding screening
5. male or non-pregnant female patients aged 18 to 80 years
6. confirmed valid health insurance

all inclusion criteria must be met

Exclusion Criteria:

1. pregnancy or breast-feeding
2. diagnosis of segmental, mixed, unclassified or undefined vitiligo
3. hypersensitivity to simvastatin or atorvastatin
4. any statins use within 8 weeks preceding eligibility screening
5. systemic immunosuppressive/immunomodulating i.e. cyclosporine A, corticosteroids within 4 weeks preceding eligibility screening or azathioprine, methotrexate, mycophenolate mofetil, Janus kinase - JAK within 8 weeks preceding eligibility screening
6. phototherapy due to vitiligo or any other medical conditions within the 4-week period preceding eligibility screening
7. any topical or systemic additional vitiligo treatment (e.g. antioxidants, ginkgo biloba, dermo-cosmetics) within 4 weeks preceding screening
8. surgical treatment of vitiligous lesions within past 4 weeks
9. hypersensitivity to statins
10. decompensated autoimmune or internal diseases
11. alcohol or drug abuse
12. skin malignancies (currently or history of skin malignancy within 5 years preceding screening)
13. presence of skin characteristics that may interfere with study assessments
14. patients currently participating in any other clinical study
15. uncooperative patients

none of the above can be met

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
evaluation of repigmentation of vitiligous lesions achieved after the administration of 1% simvastatin-acid sodium salt or 1% atorvastatin calcium salt ointments compared to vehicle ointments after a 12-week study period. | 12 weeks
  change from baseline in repigmentation on BSA and VASI scale at 12 weeks

SECONDARY OUTCOMES:
number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 weeks
  number of adverse events and serious adverse events associated with treatment
percentage of patients who achieved particular response rate as follows none 0%; poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% in each arm assessed as a relative reduction in lesional skin area | 12 weeks
  number of: poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% responders in each arm assessed as a relative reduction in lesional skin area (in sqare centimeters)
percentage of patients who achieved particular response rate as follows none 0%; poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% in each arm assessed as a relative reduction in BSA scale | 12 weeks
  number of: poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% responders in each arm assessed as a relative reduction in BSA scale
percentage of patients who achieved particular response rate as follows none 0%; poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% in each arm assessed as a relative reduction in VASI scale | 12 weeks
  number of: poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% responders in each arm assessed as a relative reduction in VASI scale
comparison of simvastatin and atorvastatin efficacy between study participants | 12 weeks
  comparison of BSA and VASI scale change between simvastatin and atorvastatin arms
the association between disease duration and repigmentation rate in study arms | 12 weeks
  the association between disease duration and repigmentation rate in study arms
the association between estimated daily ointment use (grams per square centimeter skin) and repigmentation rate | 12 weeks
  the association between estimated daily ointment use (grams per square centimeter skin) and repigmentation rate

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Czajkowski, Prof NCU, Principal Investigator — Head of Chair and Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University in Torun, Ludwik Rydygier Medical College in Bydgoszcz
Locations (1):
- Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University, Faculty of Medicine in Bydgoszcz, Bydgoszcz, Cuiavian-Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niezgoda A, Winnicki A, Krysinski J, Niezgoda P, Nowowiejska L, Czajkowski R. Topical application of simvastatin acid sodium salt and atorvastatin calcium salt in vitiligo patients. Results of the randomized, double-blind EVRAAS pilot study. Sci Rep. 2024 Jun 25;14(1):14612. doi: 10.1038/s41598-024-65722-w. PMID 38918590
- [Derived] Niezgoda A, Winnicki A, Kosmalski T, Kowaliszyn B, Krysinski J, Czajkowski R. The Evaluation of Vitiligous lesions Repigmentation after the Administration of Atorvastatin calcium salt and Simvastatin-acid sodium salt in patients with active vitiligo (EVRAAS), a pilot study: study protocol for a randomized controlled trial. Trials. 2019 Jan 25;20(1):78. doi: 10.1186/s13063-018-3168-4. PMID 30683146